CLINICAL TRIAL: NCT03991117
Title: Muscle Fibre Activation is Unaffected by Load and Repetition Duration When Resistance Exercise is Performed to Task Failure
Brief Title: Lower and Higher Load Resistance Exercise Protocols: Acute Muscle Activation and Skeletal Muscle Hypertrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Tier 1 Canada Research Chair and Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HIREB 0802
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Muscle Hypertrophy; Muscle Fibre Activation
Keywords: muscle fibre activation; electromyography
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Each individual performed four bouts of resistance exercise that varied in load and speed of contraction on two separate days (one condition each leg per visit).
Who Masked: Outcomes Assessor
Masking Description: The study investigators that performed the histochemical analysis were masked to which participant and which condition they were assessing at the time of analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 80 %1RM, Regular Tempo (Experimental): Participants performed three sets of unilateral knee extension with a load that was 80 % of their one-repetition maximum (1RM) at a tempo of three seconds per repetition.
  Interventions: Behavioral: resistance exercise
- 80 %1RM, Slow Tempo (Experimental): Participants performed three sets of unilateral knee extension with a load that was 80 % of their one-repetition maximum (1RM) at a tempo of seven seconds per repetition.
  Interventions: Behavioral: resistance exercise
- 30 %1RM, Regular Tempo (Experimental): Participants performed three sets of unilateral knee extension with a load that was 30 % of their one-repetition maximum (1RM) at a tempo of three seconds per repetition.
  Interventions: Behavioral: resistance exercise
- 30 %1RM, Slow Tempo (Experimental): Participants performed three sets of unilateral knee extension with a load that was 30 % of their one-repetition maximum (1RM) at a tempo of seven seconds per repetition.
  Interventions: Behavioral: resistance exercise

INTERVENTIONS:
Behavioral: resistance exercise — unilateral knee extensions until fatigue with varying load and speeds of contraction

SUMMARY:
How much weight an individual lifts per workout does not dictate the relative increase in muscle size the individual gains following weeks of training, which is contrary to current strength training dogma. Specifically, researchers have concluded that so long as an individual performs resistance exercise with maximum effort, it is not necessary to lift with relatively heavy loads. However, other laboratories, on the basis of surface electromyography measurements, have challenged the thesis that lighter loads can result in the hypertrophy of larger, type II muscle fibres. Therefore, the purpose of this study was to combine surface electromyography measurements with direct measurements of muscle fibre activation to see if muscle fibre activation was truly dependent on load. The investigators hypothesized that all muscle fibres would be activated when the resistance exercise was performed with maximal effort.

DETAILED DESCRIPTION:
PROCEDURES INVOLVED IN THE RESEARCH

The total time commitment of this study will be ~7 hours. Each participant's first visit (familiarization) will include an interview through where the researchers will determine if there are any reasons that the participant cannot take part in the study. The researchers will explain the study protocol and, upon the participant's consent, the investigators will obtain the participant's knee extension maximum voluntary contraction (MVC) on a dynamometer (Biodex, Shirley, USA) and a 1 repetition-maximum (RM) test on a knee extension machine. Following that, the investigators will determine the next two dates (trial days) in which the participant will come in.

The participant will be asked to come in fasted on two separate trial days, each separated by two weeks, after the participant's familiarization visit. The participant will be required to avoid physical activity 48 hours before each of the three visits. There are four conditions in this study, each varying in relative load and speed of contraction. The participant will complete two conditions on each trial day, one with each leg. The conditions include: 80%RM Normal (80N; 1 eccentric: 1 pause: 1 concentric), 80% Slow (80S; 3:1:3), 30% Normal (30N; 1:1:1) and 30% Slow (30S; 3:1:3). Each condition will include three sets to voluntary failure on a knee extension machine. Before and after each set the participant will perform three MVCs on the dynamometer identical to what the participant did on the familiarization day. The investigators will record the participant's rating of perceived exertion and effort via the Borg scale and electromyography (EMG), respectively. The participant will have one biopsy taken pre-training and two, one per condition/leg, one hour post-training.

The REB Project Number for this study is: 802

ELIGIBILITY:
Inclusion Criteria:

* healthy
* male
* 18-30 years of age

Exclusion Criteria:

* Have any acute or chronic illness such as cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin- or non-insulin dependent diabetes or other metabolic disorders-all ascertained through a medical history screening questionnaire
* Experience arthritic conditions
* Smoke tobacco products
* Consume any analgesic or anti-inflammatory drug(s), prescription or non-prescription, chronically
* Have a history of neuromuscular complications
* Are on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* Have an extensive history of RE training in the year prior to study entry.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Concentration of glycogen in muscle fibres | three weeks
  Histochemical assessment of muscle glycogen via muscle biopsies
Amplitude of electrical activity above the quadriceps muscles | three weeks
  Surface electromyography assessment via electrodes during the unilateral resistance exercise

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, PhD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to other researchers.